CLINICAL TRIAL: NCT06510010
Title: Perioperative Oxaliplatin With S-1 Combined H. Pylori Eradication in the Management of Locally Advanced Adenocarcinoma of the Gastric and Oesophagogastric Junction: an Open-label, Prospective, Multicenter, Randomised, Phase 2 Trial.
Brief Title: Perioperative Oxaliplatin With S-1 Combined H. Pylori Eradication in the Management of Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-340
Record Dates: First submitted 2024-07-11; First posted 2024-07-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy Effect
Keywords: H. Pylori Eradication; Perioperative chemotherapy; Locally Advanced Gastric Cancer
MeSH Terms: interventions — Oxaliplatin; S 1 (combination); Amoxicillin; Clarithromycin; Omeprazole; bismuth tripotassium dicitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxaliplatin With S-1 （SOX）Combined H. Pylori Eradication (Experimental): Subjects randomized to the trial group will receive 3-4 cycles of Oxaliplatin With S-1 （SOX）+ H. pylori eradication (a 14-day quadruple regimen: amoxicillin + clarithromycin + omeprazole + bismuth potassium citrate) before surgery. One of the SOX regimens will be every 3 weeks (Q3W), with a tumor response assessment at the end of the neoadjuvant therapy course. Patients will continue to receive 4-5 cycles of SOX adjuvant chemotherapy after surgery for a total of 8 cycles of SOX regimen treatment. Patients in the trial group will undergo H. pylori eradication at the time of the first cycle of the SOX regimen. H. pylori eradication will be determined by postoperative pathology, and those who are H. pylori-positive by postoperative pathology will be treated with remedial eradication therapy after recovery from surgery (except for patients with total gastric resection).
  Interventions: Drug: Oxaliplatin With S-1 (SOX) Combined H. Pylori Eradication (Amoxicillin + clarithromycin + omeprazole + colloidal bismuth subcitrate)
- Oxaliplatin With S-1 （SOX） (Active Comparator): Subjects randomized to the control group will receive 3-4 cycles of neoadjuvant therapy with the Oxaliplatin With S-1（SOX）regimen before surgery. The SOX regimen will be administered every 3 weeks (Q3W). A tumor response assessment will be performed at the end of the treatment course. Control patients were treated with H. Pylori eradication after recovery from surgery based on postoperative pathologic H. Pylori results: if H. Pylori-positive, they received H. Pylori eradication plus 4-5 cycles of SOX adjuvant chemotherapy (except for patients who underwent total gastric resection); if H. Pylori-negative, they received 4-5 cycles of SOX adjuvant chemotherapy only.
  Interventions: Drug: Oxaliplatin With S-1 （SOX）

INTERVENTIONS:
Drug: Oxaliplatin With S-1 (SOX) Combined H. Pylori Eradication (Amoxicillin + clarithromycin + omeprazole + colloidal bismuth subcitrate) — Oxaliplatin With S-1 (SOX) regimen:
  S-1: 40mg/m2, oral, bid, D1-14, one cycle every 3 weeks; Oxaliplatin: 130 mg/m2, IV, qd, D1, every 3 weeks for one cycle.
  H. pylori eradication regimen:
  H. pylori eradication was performed using a quadruple regimen for 14 d. Omeprazole 20 mg bid+Colloidal bismuth subcitrate 220mg bid+Amoxicillin 1g bid+Clarithromycin 500mg bid.
  Other Names: SOX Combined H. Pylori eradication
  Arms: Oxaliplatin With S-1 （SOX）Combined H. Pylori Eradication
Drug: Oxaliplatin With S-1 （SOX） — Oxaliplatin With S-1 （SOX） regimen:
  S-1: 40mg/m2, oral, bid, D1-14, one cycle every 3 weeks; Oxaliplatin: 130 mg/m2, IV, qd, D1, every 3 weeks for one cycle.
  Other Names: SOX
  Arms: Oxaliplatin With S-1 （SOX）

SUMMARY:
This study focuses on patients with H. pylori-positive resectable locally advanced adenocarcinoma of the gastric and oesophagogastric junction. It evaluates the perioperative oxaliplatin with S-1 (SOX) combined H. pylori eradication versus oxaliplatin with S-1 in the management of H. pylori-positive locally advanced adenocarcinoma of the gastric and oesophagogastric junction (cT3/4a Nx or T2 N2/3, M0) , assessing their values and advantages.

DETAILED DESCRIPTION:
Subjects randomized to the trial group will receive 3-4 cycles of oxaliplatin with S-1 (SOX)+ H. pylori eradication (a 14-day quadruple regimen: amoxicillin + clarithromycin + omeprazole + bismuth potassium citrate) before surgery. One of the SOX regimens will be every 3 weeks (Q3W), with a tumor response assessment at the end of the neoadjuvant therapy course. Patients will continue to receive 4-5 cycles of SOX adjuvant chemotherapy after surgery for a total of 8 cycles of SOX regimen treatment. Patients in the trial group will undergo H. pylori eradication at the time of the first cycle of the SOX regimen. H. pylori eradication will be determined by postoperative pathology, and those who are H. pylori-positive by postoperative pathology will be treated with remedial eradication therapy after recovery from surgery (except for patients with total gastric resection).

Subjects randomized to the control group will receive 3-4 cycles of neoadjuvant therapy with the SOX regimen before surgery. The SOX regimen will be administered every 3 weeks (Q3W). A tumor response assessment will be performed at the end of the treatment course. Control patients were treated with H. pylori eradication after recovery from surgery based on postoperative pathologic H. pylori results: if H. pylori-positive, they received H. pylori eradication plus 4-5 cycles of SOX adjuvant chemotherapy (except for patients who underwent total gastric resection); if H. pylori-negative, they received 4-5 cycles of SOX adjuvant chemotherapy only.

ELIGIBILITY:
Inclusion Criteria:

1. have been fully informed about the study and voluntarily signed the informed consent form (ICF);
2. Gastroscopy pathology confirmed locally advanced adenocarcinoma of the gastric and oesophagogastric junction (Siewert type I-III);
3. Clinical (enhanced CT, enhanced MRI, or PET-CT) staging at the time of diagnosis: cT3/4a Nx or T2 N2/3, M0 (The American Joint Committee on Cancer 8th edition):
4. The present H. Pylori infection at the time of diagnosis is determined by one of the following 3 items: ① Positive gastric mucosal tissue rapid urease test (RUT), tissue section staining, or bacterial culture for any of the 3 items. Positive 13C or 14C-urea breath test (UBT). ③ Positive helicobacter pylori stool antigen (HpSA) tests (clinically validated monoclonal antibody method). Positive serum H. Pylori antibody test (clinically proven reagent with high accuracy) suggests previous infection, and those who have never been treated can be considered as having current infection;
5. Sex is not limited and age is 18-75 years old;
6. Eastern Cooperative Oncology Group (ECOG) score 0-1;
7. Organ function permits major abdominal surgery;
8. Expected survival ≥ 6 months;
9. Laboratory test values must meet the following criteria within 7 days prior to enrollment:

   1. whole-body cryotherapy/cryostimulation (WBC) > 4.0 × 10^9/L and < 15 × 10^9/L, ANC > 1.5 × 10^9/L, Hb ≥ 75 g/L, PLT ≥ 100 × 10^9/L;
   2. Serum bilirubin ≤ 1.5 x high limit of normal, aspartate transaminase (AST), alanine aminotransferase (ALT) ≤ 2.5 x high limit of normal;
   3. Creatinine ≤ 1.5 x high limit of normal or creatinine clearance rate > 60 ml/min;
   4. international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × Upper limit of normal ( ULN ) only for subjects not receiving anticoagulation; subjects receiving anticoagulation should be on a stable dose;
10. Ability to cooperate with the appropriate endoscopic, laboratory and imaging tests for this protocol;
11. Females of childbearing potential (including females who are menopausal due to chemo-menopause or other medical reasons) must agree to use contraception for a period of at least 6 months from the time of signing the Informed Consent Form to at least 6 months after the last dose of study treatment or concomitant chemotherapy, whichever is later. Females must also agree to refrain from breastfeeding for a period of at least 6 months from the time of signing the informed consent to the time of the last administration of the study drug or concomitant chemotherapy, whichever is later; males must agree to use contraception for a period of at least 6 months from the time of administration of the test drug to the time of the last administration of the test drug or concomitant chemotherapy, whichever is later.

Exclusion Criteria:

1. Stage IV or unresectable gastric or gastroesophageal junction cancer as determined by the investigator;
2. Other active malignancies within 5 years or concurrently.
3. Patients who are preparing for or have previously received organ or bone marrow transplantation;
4. Myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥ 450 ms in men and ≥ 470 ms in women) within 6 months prior to the first dose (QTc interval is calculated by the Fridericia formula);
5. Presence of New York Heart Association (NYHA) class III-IV cardiac insufficiency or cardiac ultrasound: LVEF (left ventricular ejection fraction) < 50%;
6. Presence of active pulmonary tuberculosis by history or CT, or patients with a history of active pulmonary tuberculosis within 1 year prior to enrollment, or patients with a history of active pulmonary tuberculosis more than 1 year prior but without regular treatment;
7. Presence of a known active or suspected autoimmune disease. The exception is those who are in a stable state of that disease at the time of enrollment (not requiring systemic immunosuppression therapy);
8. Received a live vaccine within 28 days prior to the first dose; except inactivated viral vaccines for seasonal influenza;
9. Patients requiring treatment with systemic corticosteroids (> 10 mg/day prednisone efficacy dose) or other immunosuppressive drugs within 14 days prior to first dose or during the study period. However, enrollment is permitted if patients are allowed to be treated with topical topical or inhaled steroids, or adrenal hormone replacement therapy at doses ≤ 10 mg/day prednisone efficacy dose in the absence of active autoimmune disease;
10. Undergoing treatment in another clinical study or scheduled to begin treatment in this study less than 14 days from the end of treatment in the previous clinical study;
11. Known history of severe allergy to any study drug excipients;
12. known history of psychotropic pharmaceuticals abuse or drug addiction; patients who have stopped drinking alcohol can be enrolled;
13. Presence of patients with conditions that may increase the risk of study medication, or other severe, acute and chronic medical conditions that, in the judgment of the investigator, make participation in a clinical study unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
major pathological response (MPR) | Through postoperative pathology, an average of 2 week
  MPR defined as a tumor regression grade (TRG) score of 0-1; TRG 0 represents complete remission (no residual cancer cells), TRG 1 meant significant remission (residual lesions < 10%)

SECONDARY OUTCOMES:
pathological complete response (pCR) | Through postoperative pathology, an average of 2 week
  pCR defined as tumor regression grade (TRG) score of 0；TRG 0 represents complete remission (no residual cancer cells)
overall survival （OS） | From date of first administration until the date of death from any cause, assessed up to 36 months"
  Overall survival （OS） refers to the time from the beginning of randomization to death from any cause.
disease-free survival (DFS) | From the date of first administration until the date of first disease recurrence or date of death from any cause, whichever came first, assessed up to 36 months.
  Disease-free survival (DFS) refers to the time from the beginning of randomization to the recurrence of the disease or death from any cause (whichever occurs first).
adverse events (AE) | From the beginning of the first neoadjuvant chemotherapy to 60 days after the last adjuvant chemotherapy
  Adverse events (AE) means all adverse medical events that occur after the subject has received the experimental medication.
serious adverse events (SAE) | From the beginning of the first neoadjuvant chemotherapy to 60 days after the last adjuvant chemotherapy
  Serious adverse events (SAE) means an adverse medical event resulting in death, life-threatening, permanent or severe disability or loss of function, the need for or prolongation of hospitalization of the subject, and congenital anomalies or birth defects after the subject has received the experimental medication.
R0 resection rate | Through postoperative pathology, an average of 2 week
  No cancer cells could be found at the cut edge of the specimen under the microscope, and no cancer cells remained either visually or microscopically; the lesion was completely removed.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Lian, Ph.D, Principal Investigator — Department of Gastrointestinal Surgery, The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital，Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No
There are no plan to make individual participant data (IPD) available to other researchers.